CLINICAL TRIAL: NCT04529980
Title: Probiotics and Antibiotic Associated Diarrhea in Pediatric Complicated Appendicitis: Prospective Controlled-Comparison Trial
Brief Title: Probiotics and Antibiotic Associated Diarrhea in Pediatric Complicated Appendicitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Health (Other)
Responsible Party: Principal Investigator, Mayra Garcia, Advance Practice Practitioner, APS Administration, Children's Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STU-2019-0802
Record Dates: First submitted 2020-08-24; First posted 2020-08-28 (Actual); Results first posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Appendicitis; Appendicitis; Perforation
Keywords: Appendicitis; Probiotics
MeSH Terms: conditions — Appendicitis | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: Those randomized to the treatment group will be given probiotic therapy until discharge, while those randomized to the placebo group will be given a placebo until discharge.
Who Masked: Participant, Care Provider
Masking Description: Patients will be randomized into two study groups using randomization and utilizing a sealed envelope randomization plan. Both the care providers and study participants (parents/LAR) will be masked from which treatment assignment the participant was randomized to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lactobacillus rhanmosus GG(LGG®) Group (Experimental): Lactobacillus rhanmosus GG(LGG®)(Culturelle) is an over the counter dietary supplement that can help to restore the balance in the gut by promoting colonization to support better digestion and immune health. As such, this dietary supplement is not reviewed and approved by the FDA. This study does not intend to investigate route of administration, dose, patient population, or other factor that significantly increases the risk (or decreases the acceptability of the risk) associated with the use of the dietary supplement. Patients in the treatment group will receive a standard dose of Lactobacillus rhamnosus GG capsule following their surgery while in the hospital until discharge.
  Interventions: Dietary Supplement: Lactobacillus rhamnosus GG (LGG) Probiotic
- Placebo Control Group (Placebo Comparator): Patients in the placebo group will receive a placebo capsule following their surgery while in the hospital until discharge.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Lactobacillus rhamnosus GG (LGG) Probiotic — Lactobacillus rhanmosus GG(LGG®)(Culturelle) is an over the counter dietary supplement that can help to restore the balance in the gut by promoting colonization to support better digestion and immune health.
  Other Names: Culturelle Probiotics Digestive Health
  Arms: Lactobacillus rhanmosus GG(LGG®) Group
Dietary Supplement: Placebo — Placebo
  Arms: Placebo Control Group

SUMMARY:
To determine the effectiveness of the use of probiotics in patients with a diagnosis of complicated appendicitis on antibiotic associated diarrhea (AAD). Probiotics are defined as live microbial organisms that when administered in sufficient amounts, can provide a protective benefit to the individual patient. The use of probiotics in a pediatric population exposed to antibiotics and gastrointestinal surgery such as an appendectomy may provide a protective effect and prevent antibiotic associated diarrhea (ADD)

DETAILED DESCRIPTION:
Appendicitis is the most common urgent surgical procedure performed on children. Approximately one third of the population end up having complicated appendicitis with evidence of peritoneal contamination and infection or abscess requiring the use of IV antibiotics and prolonged hospital stay. Antibiotic Associated Diarrhea (AAD) is a common complication seen in both outpatient and inpatient settings in approximately a third of all patients treated with antibiotics (Mantegazza, et al., 2018). In particular, pediatric patients experience ADD 11-62% of the time and can up upwards to 80% in hospitalized toddlers (Mantegazza, et al., 2018). Current literature defines AAD as three or more liquid stools per day. The causes of AAD are often related to the use of multiple antibiotics, prolonged hospital stay and gastrointestinal surgery. Antibiotics often disturb the normal enteric microbiome in the gut and allow for an increased growth of pathogens (Hojsak, 2017). AAD can occur as late as six to eight weeks after antibiotic exposure. Lactobacillus rhanmosus GG(LGG®)(Culturelle) is an over the counter dietary supplement that can help to restore the balance in the gut by promoting colonization to support better digestion and immune health.This study does not intend to investigate route of administration, dose, patient population, or other factor that significantly increases the risk (or decreases the acceptability of the risk) associated with the use of the dietary supplement.At Children's Medical Center, the investigators see over 1000 cases of appendicitis a year with approximately 1/3 of those patients being complicated appendicitis. For those requiring immediate appendectomy, the typical course of treatment include surgery, admission to the hospital for 3 to 5 days, administration of IV antibiotics while in hospital, and discharge orders for oral antibiotics to complete their treatment. The investigators propose to perform a randomized controlled trial where one group of patients will receive probiotic therapy and another group of patients does not. The investigators hypothesize patients given probiotics after a diagnosis of complicated appendicitis with immediate appendectomy who receive antibiotic treatment during their inpatient stay will decrease the overall length of stay (LOS) by 25% vs the LOS in those patients who do not receive probiotics.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a post-operative diagnosis of complicated appendicitis who undergo an immediate appendectomy.
2. Patients between the ages of 4 and 18 years of age.

Exclusion Criteria:

1. Patients diagnosed with an complicated appendicitis with deferred appendectomy or non-perforated appendicitis
2. Patients that have a history of being immunosuppressed, on immunosuppression therapy, or long-term steroid therapy within the last month.
3. Patients that have central line access.
4. Patients under 4 years of age.
5. Patients that are developmentally delayed and cannot ambulate at baseline.
6. Patients with significant past medical history.
7. Patients that are in Child Protective Services custody.
8. Patients that are incarcerated.
9. Patients that are pregnant.
10. Patients that speak languages other than English and Spanish.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 98 (Actual)
Dates: Start 2020-09-08 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mayra Garcia, APRN, CNS, Principal Investigator — Children's Health
Locations (1):
- Children's Health Children's Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Agamennone V, Krul CAM, Rijkers G, Kort R. A practical guide for probiotics applied to the case of antibiotic-associated diarrhea in The Netherlands. BMC Gastroenterol. 2018 Aug 6;18(1):103. doi: 10.1186/s12876-018-0831-x. PMID 30078376
- [Background] Bethel M. Probiotics for the prevention of pediatric antibiotic-associated diarrhea: Summary of a Cochrane review. Explore (NY). 2019 Sep-Oct;15(5):382-383. doi: 10.1016/j.explore.2019.07.001. Epub 2019 Jul 11. No abstract available. PMID 31377301
- [Background] Hayes SR, Vargas AJ. Probiotics for the Prevention of Pediatric Antibiotic-Associated Diarrhea. Explore (NY). 2016 Nov-Dec;12(6):463-466. doi: 10.1016/j.explore.2016.08.015. Epub 2016 Aug 26. PMID 27688016
- [Background] Hojsak I. Probiotics in Children: What Is the Evidence? Pediatr Gastroenterol Hepatol Nutr. 2017 Sep;20(3):139-146. doi: 10.5223/pghn.2017.20.3.139. Epub 2017 Sep 26. PMID 29026729
- [Background] Mantegazza C, Molinari P, D'Auria E, Sonnino M, Morelli L, Zuccotti GV. Probiotics and antibiotic-associated diarrhea in children: A review and new evidence on Lactobacillus rhamnosus GG during and after antibiotic treatment. Pharmacol Res. 2018 Feb;128:63-72. doi: 10.1016/j.phrs.2017.08.001. Epub 2017 Aug 19. PMID 28827186
- [Background] Szajewska H, Kolodziej M. Systematic review with meta-analysis: Lactobacillus rhamnosus GG in the prevention of antibiotic-associated diarrhoea in children and adults. Aliment Pharmacol Ther. 2015 Nov;42(10):1149-57. doi: 10.1111/apt.13404. Epub 2015 Sep 13. PMID 26365389
- See also: Wanke, M. & Szajewska, H. (2014). Probiotics for preventing healthcare-associated diarrhea in — https://doi.org/10.1016/j.pepo.2013.12.003

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lactobacillus Rhanmosus GG(LGG®) Group | Placebo Control Group
Started | 57 | 41
Completed | 53 | 40
Not Completed | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lactobacillus Rhanmosus GG(LGG®) Group | Placebo Control Group | Total
Number analyzed (Participants) | 53 | 40 | 93
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 53 | 40 | 93
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.23 (3.51) | 10.53 (3.94) | 10.29 (3.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 23 | 43
  Male | 33 | 17 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 36 | 29 | 65
  Not Hispanic or Latino | 16 | 11 | 27
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 45 | 38 | 83
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 53 | 40 | 93

OUTCOME MEASURES:

1. Primary Outcome: Length of Hospital Stay
Description: Length of hospital stay measured in hours from admission to discharge. from admission to discharge, up to 1 month
Time Frame: From admission to discharge, up to 1 month
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Lactobacillus Rhanmosus GG(LGG®) Group | Placebo Control Group
Number analyzed (Participants) | 53. | 40
hours | 121.55 (59.21) | 131.69 (74.27)

2. Secondary Outcome: Number of Diarrhea Episodes Daily
Description: Documented number of diarrhea episodes each day in EHR.
Time Frame: up to 1 month
Measure: Mean (Standard Deviation); unit: episodes/day
Arm/Group | Lactobacillus Rhanmosus GG(LGG®) Group | Placebo Control Group
Number analyzed (Participants) | 53 | 40
episodes/day | 12.43 (15.51) | 9.50 (11.05)

ADVERSE EVENTS:
Time Frame: through study completion, an average of 1 month
Arm/Group | Lactobacillus Rhanmosus GG(LGG®) Group | Placebo Control Group
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/40
Other Adverse Events (participants affected / at risk) | 0/53 | 0/40

LIMITATIONS AND CAVEATS:
1. Data was pulled from documentation in the electronic medical record with the potential for missing documentation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-15): https://cdn.clinicaltrials.gov/large-docs/80/NCT04529980/Prot_SAP_001.pdf